CLINICAL TRIAL: NCT01174524
Title: Improvement of Quality of Life in Patients Using Low-dose Pills in the Different Phases of Menacme
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Geral de Fortaleza (Other Government)
Collaborators: Medley S∕A Indústria Farmacêutica (Unknown)
Responsible Party: Joao Marcos de Meneses e Silva, MD, Public Health Master, PhD Student, Hospital Geral de Fortaleza
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedleyHGF
Record Dates: First submitted 2008-12-29; First posted 2010-08-03 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2009-01

CONDITIONS: Quality of Life; Menopause; Contraception
Keywords: Quality of life; Menopause; Contraception
MeSH Terms: interventions — Gestodene; Contraceptives, Oral; Quality of Life; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gestoden and ethinylestradiol (Experimental): Gestoden 60 mcg plus ethinylestradiol 15 mcg, once a day, administered in 24∕4 regimen, for three months.
  The use of gestoden and ethinylestradiol can do an improvement of the quality of life before and after the use of the drug.Numerous large clinical trials have shown that this combination is as effective in preventing pregnancies as other oral contraceptives presently on the market. Irregular bleeding and spotting rates appear to be at least as good as older formulations. In general, the incidence of side effects associated with the progestin and estrogen components tends to be low, with very little impact on lipid and carbohydrate metabolism. . For this, the regimen can ameliorate the quality of life of the patients.
  Interventions: Drug: gestoden 60 mcg; Drug: ethinylestradiol 15 mcg

INTERVENTIONS:
Drug: gestoden 60 mcg — gestoden 60 mcg, once a day, administered in 24/4 regimen.
  Other Names: oral contraceptives; quality of life; gestodene and ethinyl estradiol
Drug: ethinylestradiol 15 mcg — ethinylestradiol 15 mcg, once a day, administered in 24/4 regimen
  Other Names: gestodene and ethinyl estradiol; quality of life; oral contraceptives

SUMMARY:
The purpose of this study is to determine whether low-dose contraceptive pills are effective in the improvement of quality of life in patients in the different phases of menacme.

ELIGIBILITY:
Inclusion Criteria:

* Fertile women with indication of use of contraceptive pills

Exclusion Criteria:

* Fertile women with any surgical contraceptive method
* Women in menopause
* Diseases the forbidden the use of the drug

Ages: 15 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Quality of life | eleven months

SECONDARY OUTCOMES:
Quality of life in differents phases of menacme | eleven months

CONTACTS AND LOCATIONS:
Overall Officials: joao MM Silva, PhD Student, Principal Investigator — Hospital Geral de Fortaleza
Locations (1):
- Hospital Geral de Fortaleza, Fortaleza, Ceará, Brazil